CLINICAL TRIAL: NCT03140878
Title: Defining the Normal Human Response to Probiotics and Developing an in Vitro System to Identify New Microbes With Probiotic Functions
Brief Title: Defining the Normal Human Response to Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Collaborators: University of Copenhagen (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HND-GI-024; H-17002470 (Registry Identifier: Regional ethical committee Denmark)
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Healthy Response to Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGG (Experimental): Lactobacillus rhamnosous (LGG) 450 billion CFU dissolved in water
  Interventions: Dietary Supplement: LGG
- Placebo (Placebo Comparator): The placebo product is the same vegetable capsule as the experimental product, identical in composition, taste and appearance but without probiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LGG — LGG is dissolved in water and consumed at one occasion (either at visit 2 or 3)
  Arms: LGG
Dietary Supplement: Placebo — Placebo is dissolved in water and consumed at one occasion (either at visit 2 or 3)
  Arms: Placebo

SUMMARY:
The study is a mono-center, randomized, semi-blinded, placebo-controlled, cross-over, proof-of principle study in healthy volunteers. The study will determine the probiotic effect of LGG on intestinal tissue and intestinal cells

DETAILED DESCRIPTION:
The study includes 3 visits. The first visit serves to check inclusion/exclusion criteria/complete questionnaire/give information about the study and receive consent. At visit 2 and 3 the included individuals will drink a placebo blend or a drink containing Lactobacillus rhamnosus GG (LGG®) and they will subsequently be biopsied from the upper intestine during endoscopy while under nurse administered propofol sedation (NAPS). There will be four weeks between visit 2 and 3.

At visit 2 and 3, biopsies will be taken from duodenum and jejunum, and luminal fluids will be collected, and one blood sample will be collected.

The down stream analysis will include a combination of gene expression analysis, microbiome analysis and classification of the individuals based on analysis of blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women
2. No medication
3. Age between 18 and 35 years
4. BMI below 30
5. Provided voluntary written informed consent

Exclusion Criteria:

1. All clinical diagnoses and disorders requiring medicine
2. Patient diagnosed with inflammatory bowel disease such as ulcerative colitis and Crohn's disease, colorectal cancer or suffering from irritable bowel syndrome.
3. Pregnant and women who are breast-feeding
4. Patient with known blood clothing disorders
5. Patients with clinical psychiatric diagnoses (including dementia)
6. Individuals who have undergone abdominal surgery, which might have effect on the GI function, except appendectomy and cholecystectomy
7. Individuals with high blood pressure (≥140 mmHg /90 mmHg)
8. Systemic use of antibiotics or steroids or antimicrobial medication in the last 4 months
9. Daily usage of NSAID in the last 2 months or incidental use in the last 2 weeks prior to screening
10. Usage of medications, except oral contraceptives, during the 14 days prior to screening
11. Lactose intolerance
12. Participation in other clinical trials in the past three months
13. Regular use of probiotics in the last 6 weeks
14. Smoking
15. Planned changes to current diet or exercise regime
16. Use of laxatives, anti-diarrheals, anti-cholinergics within last 4 weeks prior to screening
17. Use of immunosuppressant drugs within last 4 weeks prior to screening
18. Ulcer or malignancy in the intestine which is discovered during second visit

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-16 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-06-11 (Actual)

PRIMARY OUTCOMES:
Genome-wide gene expression | 3 years
  The effect of LGG on genome-wide gene expression in intestinal tissue and cells

SECONDARY OUTCOMES:
16S analysis of luminal fluid | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bornholdt J, Broholm C, Chen Y, Rago A, Sloth S, Hendel J, Melsaether C, Muller CV, Juul Nielsen M, Strickertsson J, Engelholm L, Vitting-Seerup K, Jensen KB, Baker A, Sandelin A. Personalized B cell response to the Lactobacillus rhamnosus GG probiotic in healthy human subjects: a randomized trial. Gut Microbes. 2020 Nov 9;12(1):1-14. doi: 10.1080/19490976.2020.1854639. PMID 33274667